CLINICAL TRIAL: NCT02684175
Title: Comparison of Patient & Provider Outcomes With In-Person Versus Remote Cochlear Implant Candidacy Evaluations
Brief Title: Comparison of In-Person Versus Remote Cochlear Implant Candidacy Evaluations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Bush, MD (Other)
Responsible Party: Sponsor-Investigator, Matthew Bush, MD, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-0572-P2H
Record Dates: First submitted 2016-02-06; First posted 2016-02-17 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Hearing Loss; Hearing Disorders
Keywords: Audiometry; Cochlear Implants; Adult; Telemedicine; Health Services Accessibility; Rural Population; Technology Assessment, Biomedical
MeSH Terms: conditions — Hearing Loss; Hearing Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person CI Counseling Session (Active Comparator): Participants (n=6) randomized to receive an in-person CI counseling session will receive what normally occurs with patients pursuing cochlear implantation. The counseling will last 30-45 minutes and consists 5 key components: an explanation of the patient's hearing testing results, a discussion of the impact of hearing loss on the patient's life, treatment options for hearing loss including hearing aid amplification and cochlear implantation, an explanation of how CIs function and the necessary steps in candidacy and rehabilitation, and an outline of the expected outcomes following cochlear implantation.
  Interventions: Other: In-Person CI Counseling
- Remote CI Counseling Session (Experimental): Participants (n=6) randomized to receive a remote CI counseling session will be receiving the counseling session remotely. The participants will be counseled remotely by the audiologist located in Lexington, KY via the telemedicine system (intervention). This counseling will last 30-45 minutes and consists 5 key components: an explanation of the patient's hearing testing results, a discussion of the impact of hearing loss on the patient's life, treatment options for hearing loss including hearing aid amplification and cochlear implantation, explanation of how CIs function and the necessary steps in candidacy and rehabilitation, and an outline of the expected outcomes following cochlear implantation.
  Interventions: Device: Remote CI Counseling

INTERVENTIONS:
Device: Remote CI Counseling — The remote setup includes a 500 series teleconference audio and video live set-up. The teleconference set-up will be situated on a telemedicine cart and placed within the sound-proof booth at the testing site (UK ENT practice in Morehead, KY). The audiologist will deliver the session remotely.
  Other Names: Polycom 500 series
  Arms: Remote CI Counseling Session
Other: In-Person CI Counseling — The standard face-to-face counseling that will occur between the participant and audiologist is the standard of care. No technology will be used. The audiologist will deliver the session face-to-face with the participant in the same room (standard practice).
  Arms: In-Person CI Counseling Session

SUMMARY:
The objective of this study is to compare remote and in-person audiological cochlear implant candidacy evaluations (including audiological (hearing) testing and counseling sessions) in a rural Appalachian region.

DETAILED DESCRIPTION:
In Aim 1, participants (N=42) will receive both an in-person (standard of care) and remote (experimental) comprehensive audiological evaluation.Participants will be randomized to receive both sessions in a particular sequence (in-person, remote versus remote, in-person) to reduce order effect. Remote audiological sessions will involve face-to-face communication and testing over a high-speed hard wired connection (10 Mgb/s) conducted within the University of Kentucky firewall protection using a Polycom 500 series teleconference audio and live video set-up. The audiologist will direct the remote audiological evaluation with the participant (in the UK Otolaryngology (ENT) practice in Morehead, KY) from a work station at the Otolaryngology (ENT) practice in Lexington, KY. Evaluations will include pure-tone air and bone conduction thresholds (level of hearing ability) along with speech audiometry (speech recognition thresholds and word recognition scores). Scores from the Arizona Biological (AzBio) test (speech recognition) completed remotely and in-person will be compared for each person to determine equivalence. Upon enrollment, participants will fill out a demographic questionnaire along with an adapted version of the University of Rhode Island Change Assessment (URICA) questionnaire, assessing their current stage of change toward seeking hearing rehabilitation.

Aim 2 will involve participants from Aim 1 (N=12). Half of the cohort (n=6) will be randomized to receive a remote cochlear implant counseling session (experimental) and the other half (n=6) will be randomized to receive an in-person cochlear implant counseling session (standard of care). Both sessions will occur in the ENT practice in Morehead, KY with an audiologist but the audiologist will be physically located in the ENT practice in Lexington, KY directing the session during the remote sessions. The counseling session lasts 30-45 minutes and consists of 5 key components: an explanation of the patient's hearing testing results, a discussion of the impact of hearing loss on the patient's life, treatment options for hearing loss including hearing aid amplification and cochlear implantation, an explanation of how cochlear implants function and the necessary steps in candidacy and rehabilitation, and an outline of the expected outcomes following cochlear implantation. After participants receive either remote or in-person session, they will complete a satisfaction questionnaire on the session and the URICA questionnaire.The URICA questionnaire is a validated assessment tool measuring an individuals' motivation for change by providing a score that places them within one of the four categories: precontemplation, contemplation, action and maintenance (Laplante-Lavesque, Hickson, & Worral, 2013). After each session, the audiologist will fill out a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>18) who are current patients at the University of Kentucky Morehead Clinic
2. Adults who have moderate to profound hearing loss
3. Adults who can speak and understand English since cochlear implantation candidacy testing is performed using standardized word lists in English

Exclusion Criteria:

1. Adults with prelingual deafness
2. Adults who use sign language as a primary means of communication
3. Adults with active otological infections with otorrhea or cerumen impaction seen on otoscopy
4. Pregnant women since pregnant women are not cochlear implant surgical candidates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
(Aim 1): Comparison of Remote Audiological Testing Scores with In-Person Audiological Testing Scores | 2 weeks
  Arizona Biological (AzBio) scores gathered remotely via the telemedicine system will be compared to AzBio scores gathered via in-person (face-to-face) per participant.
(Aim 2): Remote Cochlear Implant Counseling Completion Rate | 45 minutes
  The number of participants that enroll into Aim 2 will be recorded and compared to the number of participants that complete all study-related activities within this Aim.
(Aim 2): In-Person Cochlear Implant Counseling Participant Feedback | 10 minutes
  Participants in Aim 2 that receive an in-person session will complete a 6-question satisfaction questionnaire post cochlear implant counseling session.
(Aim 2): In-Person Cochlear Implant Counseling Provider Feedback | 10 minutes
  Provider(s) in Aim 2 that deliver in-person session(s) will complete a 6-question satisfaction questionnaire post cochlear implant counseling session.
(Aim 2): Remote Cochlear Implant Counseling Participant Feedback | 10 minutes
  Participants in Aim 2 that receive a remote session will complete a 13-question satisfaction questionnaire post cochlear implant counseling session.
(Aim 2): Remote Cochlear Implant Counseling Provider Feedback | 10 minutes
  Provider(s) in Aim 2 that deliver remote session(s) will complete a 13-question satisfaction questionnaire post cochlear implant counseling session.
(Aim 2): Stage of Change toward Seeking Hearing Rehabilitation | 2-4 weeks
  Participants in Aim 2 will complete the University of Rhode Island (URICA) questionnaire post cochlear implant counseling session. This questionnaire will determine the participant's stage of change toward seeking hearing rehabilitation. These URICA scores will be compared to URICA scores gathered in Aim 1 for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Bush, MD, Principal Investigator — University of Kentucky Department of Otolaryngology - Head & Neck Surgery
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laplante-Levesque A, Hickson L, Worrall L. Stages of change in adults with acquired hearing impairment seeking help for the first time: application of the transtheoretical model in audiologic rehabilitation. Ear Hear. 2013 Jul-Aug;34(4):447-57. doi: 10.1097/AUD.0b013e3182772c49. PMID 23364333
- [Result] Fletcher KT, Dicken FW, Adkins MM, Cline TA, McNulty BN, Shinn JB, Bush ML. Audiology Telemedicine Evaluations: Potential Expanded Applications. Otolaryngol Head Neck Surg. 2019 Jul;161(1):63-66. doi: 10.1177/0194599819835541. Epub 2019 Mar 5. PMID 30832542